CLINICAL TRIAL: NCT06193408
Title: Assessment of a Novel Fixed-dose Combination (FDC) Drug VR-AD-1005 for the Treatment of Acute Watery Diarrhea in Cholera: a Phase II, Randomized, Placebo-controlled, Double-blinded Efficacy and Safety Trial
Brief Title: Assessment of a Novel Fixed-dose Combination (FDC) Drug VR-AD-1005 for the Treatment of Acute Watery Diarrhea in Cholera
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunazine Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-23089
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: randomized, placebo-controlled, double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR-AD-1005 (Experimental)
  Interventions: Drug: VR-AD-1005
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VR-AD-1005 — oral capsule
  Arms: VR-AD-1005
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
Cholera still remains a global public health concern affecting both children and adults, and patients can succumb in quick time if remain untreated. Cholera is a secretory diarrhea and is generally treated with oral or intravenous rehydration therapy to compensate for the fluid loss. However, antimicrobial treatment is given to patients with moderate to severe diarrhea. The consistent emergence of multidrug-resistant bacteria is a major concern for the management of infectious diseases including cholera. No antisecretory drug has so far been proven successful. In a phase II clinical trial, the investigators will assess the effectiveness of a novel antisecretory drug VR-AD-1005 for treating cholera. Changes in stool volume and rehydration therapy will be assessed for VR-AD-1005 in comparison with placebo. If successful, this will be a huge advance in managing cholera and other secretory diarrhea. The introduction of the antisecretory drug can minimize the hospital stay and reduce antibiotic use, which in turn can reduce the emergence of antibiotic resistance among pathogens

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Adults, both genders aged 18-65 years.
* Acute watery diarrhea (defined as passage of three or more liquid stools within the 24 hours before admission) with severe dehydration on arrival.
* Detection of V. cholerae by rapid diagnostic assay (e.g. dark field microscopy).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Subjects with passage of bloody stools or muco-purulent stools.
* Subjects with chronic diarrhea (>4 weeks of Diarrhea).
* Clinically significant concomitant systemic disease (i.e. cardiovascular diseases including heart failure, acute kidney injury, sepsis or life-threatening malignant cancer).
* Mental incapacity, unwillingness, or language barriers, precluding adequate understanding or cooperation.
* History of receiving antimicrobial or antidiarrheal drugs within 6 hours prior to admission.
* Positive urine pregnancy test for all female patients
* Failure to obtain informed consent.
* Failure to definitively diagnose cholera via culture or RT-PCR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Change in stool output volume during treatment period. | 3 days
  Change in stool output volume (ml/hour) over a treatment period measured and plotted as total stool output during 12-hour stool collection at every 12 hours for 72 hours

SECONDARY OUTCOMES:
Time until the stool volume output of 200 ml/hour | 3 days
  time (hours) from start of treatment until the stool output changes (reduces) to 200 ml/hour or less
Number of subjects with clinical recovery | 3 days
  Total number of subjects achieving clinical recovery during treatment period expressed as a fraction of the total subjects per treatment arm.
Number of unscheduled IV rehydration episodes per treatment | 3 days
  Average number of unscheduled IV rehydration episodes per participant per treatment arm.
Duration of IV rehydration | 3 days
  Average duration of IV rehydration per subject per treatment arm expressed in hours.
Adverse Events Occurrence | 28 days
  Average number of adverse events per subject per treatment arm

CONTACTS AND LOCATIONS:
Locations (1):
- Icddr,b, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No